CLINICAL TRIAL: NCT05974007
Title: Neoadjuvant Treatment Real-world Clinical Outcomes in NSCLC: A Retrospective Multi-center Study (NeoR-World)
Brief Title: Neoadjuvant Treatment Real-world Clinical Outcomes in NSCLC
Acronym: NeoR-World
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 22/093-3294
Record Dates: First submitted 2023-07-19; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Neoadjuvant immunochemotherapy; Neoadjuvant chemotherapy; Real world study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Resectable stage I-III NSCLC: Patients with NSCLC patients receiving neoadjuvant therapy and undergoing surgeries. Resectability after neoadjuvant therapy is judged by the multidisciplinary team of thoracic surgeon, oncologist and radiation oncologist.
  Interventions: Drug: Neoadjuvant immunochemotherapy; Drug: Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant immunochemotherapy — Patients with operable stage I-III NSCLC who have previously undergone platinum drugs and immune checkpoint inhibitors(Anti PD-1) and then undergone radical surgery
  Other Names: Neoadjuvant immunotherapy
Drug: Neoadjuvant chemotherapy — Patients with operable stage I-III NSCLC who have previously undergone platinum-based chemotherapy regimens and then undergone radical surgery
  Other Names: Neoadjuvant platinum-based doublet chemotherapy

SUMMARY:
Despite the clinical success of immune checkpoint blockade (ICB), in neoadjuvant setting, there is still a lack of valid data for operable NSCLC in the real world. This study aim to compare the clinical outcomes (pathologic response rate versus survival) of neoadjuvant immunochemotherapy with neoadjuvant chemotherapy in the real world, to explore the impact of clinicopathological factors on clinical outcomes in neoadjuvant immunochemotherapy setting, and to identify potential neoadjuvant immunochemotherapy beneficiaries.

DETAILED DESCRIPTION:
Although the application of neoadjuvant immunotherapy in NSCLC has brought a new treatment option to many patients, most evidence is based on interventional clinical trials, in which the participants are highly selected and the therapeutic strategies are restricted, resulting in limited representation. There is still a lack of large-scale multicenter real-world data to further verify the benefits in long term overall survival, identify the potential beneficiaries and optimize the therapeutic strategies of neoadjuvant immunochemotherapy.

To meet the forementioned need, the investigators will perform a multi-center retrospective cohort to describe the patterns of neoadjuvant immunochemotherapy use in real world, compare the efficacy of neoadjuvant immunochemotherapy ,and evaluate prognosis of neoadjuvant immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Cytological or histological diagnosis of non-small cell lung cancer
2. Patients who have previously undergone neoadjuvant immune checkpoint inhibitors and/or chemotherapy and then undergone radical surgery;
3. Stage I-III non-small cell lung cancer (IASLC/UICC staging eighth edition);
4. No previous history of malignant tumors and other malignant tumors at the same time, without any anti-tumor treatment;
5. ECOG score 0-1, heart, lung, liver, brain and kidney function can tolerate surgery;
6. At least one measurable lesion (RECIST v1.1);
7. Age >= 18 years old and <= 85 years old;
8. Be able to abide by the visits and related procedures stipulated in the program.

Exclusion Criteria:

1. Patients included in anti-tumor drug intervention or unblinded clinical trials, in which the treatment being administered is unknown.
2. Prior surgery, radiotherapy or systemic therapy for NSCLC, including radiofrequency ablation, etc.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stage I-III NSCLC patients undergo neoadjuvant treatment.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival(DFS) | DFS was defined as the time from surgery to the appearance of metastasis, up to approximately 5 years.
  Defined as the time from the date of randomization until the date of disease recurrence or death (by any cause in the absence of recurrence).
Pathological Complete Response (pCR) | Within 2 weeks after surgery
  defined as 0% of viable tumor cells in primary tumor and lymph nodes

SECONDARY OUTCOMES:
OS (overall survival) | From date of surgery until date of death due to any cause, up to approximately 5 years.
  OS is defined as the time from surgery tiem until death from any cause.
Overall Survival (overall survival) Rate | From date of surgery until date of death due to any cause. Assessed at 1 years.
  OS is defined as the time from surgery tiem until death from any cause, estimated from a Kaplan Meier plot of OS at the time of the primary analysis.
Overall Survival (overall survival) Rate | From date of surgery until date of death due to any cause. Assessed at 2 years.
  OS is defined as the time from surgery tiem until death from any cause, estimated from a Kaplan Meier plot of OS at the time of the primary analysis.
Overall Survival (overall survival) Rate | From date of surgery until date of death due to any cause. Assessed at 5 years.
  OS is defined as the time from surgery tiem until death from any cause, estimated from a Kaplan Meier plot of OS at the time of the primary analysis.
EFS (event-free survival) | Up to 5 years after first therapy.
  EFS was defined as time from study inclusion (first dose date) to disease progression, death, or discontinuation of treatment.
Event Free Survival (event-free survival) Rate | From date of first received neoadjuvant therapy to 1 years after neoadjuvant.
  EFS was defined as time from study inclusion (first dose date) to disease progression, death, or discontinuation of treatment.
Event Free Survival (event-free survival) Rate | From date of first received neoadjuvant therapy to 2 years after neoadjuvant.
  EFS was defined as time from study inclusion (first dose date) to disease progression, death, or discontinuation of treatment.
Event Free Survival (event-free survival) Rate | From date of first received neoadjuvant therapy to 5 years after neoadjuvant.
  EFS was defined as time from study inclusion (first dose date) to disease progression, death, or discontinuation of treatment.
Major Pathological Response (MPR) | Within 2 weeks after surgery
  defined as ≤10% of viable tumor cells
Patterns of Relapse | Within 5 years after surgery
  Relapse was defined as disease recurrence at any site.

CONTACTS AND LOCATIONS:
Overall Officials: Jie He, Dr., Study Chair — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China